CLINICAL TRIAL: NCT05844943
Title: Part II of Two-Part Early Feasibility Study to Evaluate the Safety and Tolerability of a Novel Negative Pressure Wound Therapy Glove for Hand Injuries
Brief Title: Early Feasibility Study of a Novel Negative Pressure Wound Therapy Glove for Hand Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Christopher Allan, Associate Professor, School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00017024; UL1TR002319 (NIH)
Record Dates: First submitted 2023-04-07; First posted 2023-05-06 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-01

CONDITIONS: Hand Injuries
MeSH Terms: conditions — Hand Injuries | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Soft tissue hand injury (Experimental)
  Interventions: Device: ReHeal glove with Negative Pressure Wound Therapy (NPWT)

INTERVENTIONS:
Device: ReHeal glove with Negative Pressure Wound Therapy (NPWT) — ReHeal glove hand dressing with Negative Pressure Wound Therapy (NPWT).

SUMMARY:
Single-center nonrandomized single-arm early feasibility study of participants with soft tissue trauma in the hand. Prior to enrolling participants with hand injuries, the safety of continuous glove use for up to 96 hours without a glove replacement will be assessed on healthy volunteers.

Injured participants will be on study for up to 7 weeks depending on when the final glove is removed.

Screening: Prior to surgery and through 72 hours post-surgery to identify eligible patients

Treatment with Glove: Treatment begins with initial application of the ReHeal Glove and can last up to 7 days (with dressing changes every 48-72 hours unless more frequent changes are requested by the treating physician.)

Follow-up: Up to 6 weeks after final removal of glove to ensure complete wound healing.

DETAILED DESCRIPTION:
A maximum of 10 participants may be enrolled. Each participants will be enrolled sequentially, with in-depth review of study data from each individual participant before proceeding to the next participant. There will be one and only one participant at a time experiencing glove use. This allows the study team to identify and correct any safety issues before another participant is enrolled and begins glove use. This strategy is in place to minimize risk to participants. Screening data will be reviewed to determine participant eligibility. Participants who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

Each participant will have the glove applied after surgery. The timing of the initial application could be immediately following surgery or up to 3 days after the surgery, at the discretion of the treating surgeon. Application delays of 1-3 days may be indicated if, in the opinion of the surgeon, the wound would benefit from a period of immobilization prior to donning the glove and allowing for the additional mobility possible with the glove dressing.

Reasons for a potential delay could include minimizing bleeding or oozing after debridement, or for protection of a skin graft. Following current standards of negative pressure wound therapy (NPWT), the wound will be assessed and the glove replaced every 48 to 72 hours. The glove may be assessed by the clinical care team and, if needed, removed and replaced earlier. At each participant encounter, data will be collected by the study team and pressure settings will be documented. At each study visit involving a dressing change, the glove will be removed for closer assessment of the wound and replaced with a new glove. Participants will remain in the study until wound healing or clinical resolution, or study exit. After study exit for each participant, data will be reviewed, and any design changes indicated by the results of the study will be implemented prior to enrollment of the next subject.

The ReHeal Glove and Cardinal Health Negative Pressure Wound Therapy Pro/Pro To Go pump will be used.

ELIGIBILITY:
Inclusion Criteria:

* • Persons 22 years or older

  * Wound size greater than 1cm2
  * Patient will have surgery to treat the wound, warranting the use of a dressing after surgery
  * Patient must be able to give informed consent
  * Persons who can read and write in English
  * Acute, unilateral, and isolated open finger or hand injuries caused by:

    * Burn
    * Blast
    * Abrasion
    * Avulsion
    * Amputation
    * Mangling hand injury
    * post-compartment syndrome release ((fasciotomy) and debridement
    * flexor tendon repair
    * exposed nerve or tendon
    * open wounds not yet ready for flap or graft
    * wounds after graft or flap
    * crush injuries associated with fractures (open or closed) which do not require stabilization and can therefore accommodate hand motion (for example, an abrasion injury may involve loss of some portion of cortical bone due to friction without losing structural stability sufficient to permit finger motion).
    * Fasciectomy
    * Tenolysis

Exclusion Criteria:

* • Polytrauma outside of the hand

  * Malignancy in the wound
  * Patient undergoing active chemotherapy
  * Hand wound with any untreated infection
  * Contaminated wounds not yet debrided
  * Insensate hand
  * Non-debrided tunneling wounds
  * Necrotizing soft-tissue infections
  * Osteomyelitis
  * Fractures requiring stabilization.
  * Untreated non-enteric fistulas
  * Smoker
  * Hemophiliac
  * Sepsis
  * Active cellulitis in the wound area
  * Radiation applied directly to the wound
  * Patients with allergies to product components: silicone, silicone adhesives and polyurethane films (direct contact with wounds), acrylic adhesives (direct contact with skin), polyethylene fabrics, and super-absorbent powders (polyacrylates within the dressing).
  * Patients chronically treated with any of the following medications:

    * Anti-coagulants
    * Immunosuppressants
    * Corticosteroids
    * NSAIDs

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Did significant adverse events occur | 0-7 days
  Did infection or skin injury occur
Skin remains intact | 0-7 days
  Did maceration occur.
Dressing changes | 0-7 days
  Total number of dressing changes.
Additional adverse events | 0-7 days
  Type and severity of adverse events.

SECONDARY OUTCOMES:
Hand Function (through range of motion) | 7 days to 12 weeks
  Total Active Motion of fingers
Hand Function (through range of motion) | 7 days to 12 weeks
  Opposition of thumb
Hand Function (grip and pinch strength) | 7 days to 12 weeks
  Grip and Pinch Strength
Time to healing | 7 days to 12 weeks
  Wound closure rate will be assessed by documenting wound size at each clinic visit.
Incidence of additional surgical procedure/interventions | 7 days to 12 weeks
  Where there any repeat debridement, skin grafts, flaps, or other procedures will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H Allan, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No